CLINICAL TRIAL: NCT03967028
Title: Indication of Ceaseran Section in Primigravida According to Robson's Classification
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: CSR
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: CESAREAN SECTION
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: primigravida scheduled for cesarean section
  Interventions: Procedure: cesarean section

INTERVENTIONS:
Procedure: cesarean section — lower segment cesarean section either elective or emergency

SUMMARY:
Rate of caesarean section surgery are rising worldwide,but the determinant of this increase,especially in low-income and middle-income countries, are controversial.In 1985,The world Health organization (WHO) stated;(There is no justification for any region to have a ceasearan section rate higher than 10-15%). Despite the lack of scientific evidence indicating any substantial maternal and perinatal benefits from increasing cs rates,and some studies showing that higher rates could be linked to negative consequences in maternal and child health, CS continue to increase world wide

ELIGIBILITY:
Inclusion Criteria:

* Nullipara
* Single fetus .
* More than 37 weeks .
* Patients who pass into spontaneous
* Patient who induced labour

Exclusion Criteria:

* Non cephalic presentation.
* Abnormal lie

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women admitted to women health hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The prevalence of etiologies of cesarean section | one month
  determine the rate of cesarean section with different indication according to Robson classification

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt